CLINICAL TRIAL: NCT05614648
Title: A Phase 3, Prospective, Multicenter, Randomized, Double-blind, Sham-controlled Study of the Efficacy and Safety of STX-015 in the Treatment of Pain Associated With Lumbosacral Radiculopathy
Brief Title: Sciatica Epidural Radiculopathy Experimental New Interventional TherapY Clonidine Micropellet
Acronym: SERENITY CM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Loss of funding- Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: Sollis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STX-015-23-01
Record Dates: First submitted 2022-10-27; First posted 2022-11-14 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Lumbosacral Radiculopathy

STUDY DESIGN:
Intervention Model Description: Clonidine Micropellet vs Sham-Control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Clonidine Micropellets Injection (Active Comparator): Clonidine Micropellets single dose injection into the lumbar epidural space
  Interventions: Drug: Clonidine Micropellets; Device: Tuohy epidural needle
- Sham Insertion (Sham Comparator): Sham Control non-epidural needle placement
  Interventions: Device: Tuohy epidural needle

INTERVENTIONS:
Drug: Clonidine Micropellets — 0.975 mg clonidine hydrochloride as 3 micropellets administered in one injection
  Arms: Clonidine Micropellets Injection
Device: Tuohy epidural needle — 18-gauge Tuohy epidural needle using a custom-built injector

SUMMARY:
This study will evaluate the safety and effectiveness of a new pain medication in development, clonidine micropellet. Participants will receive a single injection of either clonidine micropellet or sham injection for the treatment of low back and leg pain from sciatica.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between 18 and 70 years of age (inclusive) at time the Informed Consent Form (ICF) is signed.
2. Must have a primary diagnosis of unilateral lumbar and/or lumbosacral radiculopathy defined by all of the following: supported by history, physical examination, and radiologic pathology consistent with a disc protrusion, non-sequestered extrusion, or sequestered fragment, as evidenced by magnetic resonance imaging (MRI), that is consistent with the clinical signs and symptoms of lumbar or lumbosacral radiculopathy.
3. Subject's pain must have a radicular component (radiation into the leg along the L3-S1 [inclusive] dermatomal pattern) and may or may not be associated with additional neuropathic features such as reduced sensory, motor, or deep tendon reflexes.

   1. Worst radicular pain symptoms should be confined to a single dermatomal level as confirmed on physical examination (to allow determination of injection level).
   2. The NRS leg pain must be ≥4, must extend below the knee and be consistent with one of the dermatomal distributions noted above.
   3. Radicular pain symptoms in the current episode must have been present for at least 8 weeks, but not longer than 9 months at the time of Screening.
   4. Subjects must not have had a significant reduction in the pain in the 1 to 2 weeks before Screening (i.e., pain must not be improving significantly based on the discretion of the Investigator).
4. Baseline 0-10 NRS average pain score localized to at least 1 target location must be ≥6 and ≤9.
5. Subjects must be able to separately distinguish and characterize the contribution of back and leg pain to their overall pain to independently assess the response of each to intervention. Investigators must confirm that subjects can do so based upon pain diagrams and direct questioning.
6. Subjects must have had no significant improvement following a minimum of 8 weeks of the following categories prior to Screening:

   1. Mechanical intervention (eg, physical therapy, home exercise program, heat compresses/massage, chiropractic treatment), and
   2. Over-the-counter analgesics (non-steroidal anti-inflammatory drugs, topical patches/creams/gels/ointments).
7. Subjects of childbearing potential must have a negative (serum) pregnancy test at Screening and a negative urine pregnancy test within 24 hours before the injection procedure and must commit to either abstain continuously from sexual intercourse or to use, at the Investigator's discretion, highly effective birth control during the study period.
8. Must sign an ICF indicating that they understand the purpose and any risks associated with the procedure required for the study and is willing to participate in the study to completion.
9. Must be willing and able to adhere to the prohibitions and restrictions specified in the protocol.
10. Must be able to read, write, understand, and complete study-related tasks, and adequately communicate regularly with the site.
11. Must have an email address and access to the internet from an electronic device in order to complete daily EDQ information.

Exclusion Criteria:

1. Subject has significant pain unrelated to the lumbar or lumbosacral radiculopathy (eg, knee pain, hip pain, or rib pain) that, in the Investigator's opinion, could require chronic analgesic treatment and interfere with the assessment of IP therapeutic effect.
2. Subject has radiological findings or presenting features such as severe motor weakness (with or without reduced deep tendon reflexes) and is a candidate for surgical referral (i.e., progressive neurologic deficit or cauda equina syndrome).
3. Subject has evidence of pathology on MRI (obtained during the current episode of pain) that may result in pain unlikely to be addressed by the IP, including but not limited to the following:

   1. Symptomatic (eg, neurogenic claudication) radiographically confirmed central stenosis at any level or diffuse spine pathology.
   2. Non-inflammatory or bony lateral recess or foraminal stenosis such as that caused by facet hypertrophy or osteophytes that is a significant contributor to the current episode of pain.
   3. Spondylolisthesis > 3 mm at the level of the involved dermatome.
   4. Evidence of a lumbar vertebral compression fracture, synovial cyst, lumbar epidural lipomatosis, or extraforaminal pathology.
4. Subject has a history of, or current diagnosis of, fibromyalgia.
5. Subject has a history of lumbar surgery and/or intradiscal interventions (including discography).
6. Subject has an active infection (eg, fever or other objective evidence of an infection within 7 days of the planned injection) or any skin condition visible at the injection site at time of Screening.
7. Subject has evidence of a coagulation abnormality or history of abnormal bleeding or is on anticoagulation therapy at time of Screening.
8. Subject has current untreated or clinically significant anxiety and/or depression as defined by the following:

   1. Beck Anxiety Inventory® (BAI®) score ≥29 or,
   2. Beck Depression Inventory-2® (BDI®) score ≥31.
   3. Changes in medications administered for treatment of depression or anxiety within the 30 days before Screening. Note: If a subject is taking antidepressant or anti-anxiety medication, either for the treatment of depression/anxiety or as an analgesic adjunct, the subject must agree to maintain a stable dose (no change in dosage) for the first 3 months of the study.
9. Subject is planning to receive a spinal injection or spine procedure while participating in this study, unless this procedure can be postponed until study completion.
10. Subject has received an ESI, nerve block, or other similar procedure in the lumbosacral area performed during the 8 weeks prior to Screening.
11. Subject is receiving or has received the following medications prohibited in this study:

    1. Short-acting opioids taken as needed (PRN) less than 4 days a week (hydrocodone, oxycodone, tramadol, etc.) within 14 days prior to Screening.
    2. Long-acting opioids or short-acting opioids taken regularly, i.e., more than 4 days a week within 30 days prior to Screening.
    3. Anticonvulsants for treatment of radicular leg pain if the dose has changed in the 30 days prior to Screening or the subject is unable to maintain a stable dose for the first 3 months of the study.
    4. Systemic corticosteroids within the 30 days prior to Screening.
    5. Central alpha-agents, including clonidine-containing medication or dexmedetomidine within 30 days before Screening.
12. Subject has a history of treatment, or has been recommended for treatment, of alcohol or drug use disorder treatment within the year prior to Screening.
13. Subject has a known or suspected allergy, hypersensitivity, or intolerance to any of the following:

    1. Clonidine/clonidine hydrochloride.
    2. Polylactic acid (found in products such as Lupron Depot®, Atridox®, some types of dermal fillers, and some types of sutures).
    3. Radiographic contrast agents or any other medications to be used during the procedure.
14. Subject has recent (within previous 8 weeks) symptomatic hypotension, orthostatic hypotension, or bradycardia.
15. Subject has a Body Mass Index (BMI) or a body habitus that, in the Investigator's judgment, would require a needle longer than a 3.5-inch Tuohy needle.
16. Subject has participated in a clinical trial of an investigational drug or device within 30 days of Screening.
17. Subject has previously participated in a clinical trial sponsored by Sollis Therapeutics (including Protocol Number STX-015-18-01 and Protocol Number STX-015-18-02).
18. Subject has any medical condition that, in the Investigator's opinion, could adversely impact study participation or safety, require chronic analgesic treatment, or interfere with the pain assessments (eg, painful neuropathy, rheumatologic disorder, etc.).
19. Subject has worker's compensation benefits and/or is involved in any litigation related to his/her radicular pain.
20. Subject is currently pregnant or breast feeding, planning to become pregnant or, if of childbearing potential, is unwilling to have a pregnancy test administered or use appropriate, highly effective contraception.
21. Subject is unable or unwilling to undergo MRI examinations.
22. Subject is unable to adequately rate his/her pain in the EDQ.
23. Presence of active kidney disease, as evidenced by an estimated glomerular filtration rate of less than 60 mL/min/1.73m2 utilizing the Chronic Kidney Disease Epidemiology Collaboration equation.
24. Subjects will be excluded from randomization if they have any of the following during the 7-day Baseline Period:

    1. Two or more ratings of NRS Average Leg Pain and/or Back Pain > 9 (showing severe pain),
    2. Two or more ratings of NRS Average Leg Pain and/or Back Pain ≥ 9 AND ≤ 3 (showing inconsistent pain).
25. Employees of Sollis Therapeutics, Novotech Health Holdings, or study site personnel directly affiliated with this study, and their immediate family members. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Primary efficacy: Pain Intensity Difference (PID) for the average pain Numeric Rating Scale (NRS) from baseline to D90 in lumbosacral radiculopathy. | Baseline to day 90
  Difference in average pain score, using a scale of 0-10 with 0 no pain and 10 worst possible pain, from baseline to day 90.
Incidence of Treatment-Emergent Adverse Events. | Baseline to day 90
  Difference in incidence of adverse events and treatment due to radicular leg pain from Baseline to day 90 post injection based on physical examination findings and vital signs measurements.
Incidence of symptomatic hypotension as an adverse event of special interest. | Baseline to day 90
  Difference in incidence defined as low blood pressure associated with subject-reported symptoms of dizziness, lightheadedness, syncope, blurred vision, or nausea.

SECONDARY OUTCOMES:
Change in Oswestry Disability Index (ODI) score | Baseline to month12
  6 categories of 10 question, each question is scored from 0-5 (minimum to maximum). The scores range from 0-100% with lower scores meaning less disability.
Difference in Rescue medication consumption. | Baseline to month12
  Consumption from baseline through day 30
Change in Average and Worst NRS from Day 90 post injection to 12 months post injection. | from Day 90 to month 12 post injection
  Difference in NRS pain scores from Day 90 to month 12 post injection.
Percent of subjects with significant improvement in pain. | Baseline to day 90
  30 percent improvement in pain from baseline to day 90.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Pima Pain Center (site 125), Tucson, Arizona
  - University of Arizona/Banner (site 116), Tucson, Arizona
  - Quality of Life Medical & Research Centers, LLC (site 127), Tucson, Arizona
  - UCSD (site 124), La Jolla, California
  - Nurovations/Napa Pain Institute (site 107), Napa, California
  - International Spine, Pain & Performance Center (site 118), Washington D.C., District of Columbia
  - Mocasa Wellness Center (site 119), Miami, Florida
  - AMPM Research Clinic (site 106), Miami, Florida
  - Florida Pain Relief Group (site 126), Tampa, Florida
  - Conquest Research (site 142), Winter Park, Florida
  - Injury Care Research (site 130), Boise, Idaho
  - University of Kansas Medical Center (site 137), Kansas City, Kansas
  - Neuroscience Research Center (site 105), Overland Park, Kansas
  - Brigham and Women's Hospital (site 129), Chestnut Hill, Massachusetts
  - St. Louis Pain Consultants (site 134), Chesterfield, Missouri
  - Wake Forest Pain & Spine Specialists (site 112), Clemmons, North Carolina
  - The Center for Clinical Research (site 101), Winston-Salem, North Carolina
  - Cleveland Clinic (site 121), Cleveland, Ohio
  - University Hospitals (site 131), Cleveland, Ohio
  - Clinical Investigations LLC (site 103), Edmond, Oklahoma
  - Pacific Sports and Spine, LLC (site 133), Eugene, Oregon
  - Clinical Trials of South Carolina (site 114), Charleston, South Carolina
  - HRMD Research (site 102), Dallas, Texas
  - UT Southwestern (site 140), Dallas, Texas
  - NCP Clinical Research (site 141), Houston, Texas
  - Texas Pain Consultant Associates (site 110), Sugar Land, Texas
  - ARH Research, LLC (site 108), The Woodlands, Texas
  - Space City Pain (site 135), Webster, Texas
  - Physicians' Research Options (site 122), Draper, Utah
  - CenExel JBR Clinical Research (site 113), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No